CLINICAL TRIAL: NCT00896987
Title: An Open, Randomized, Multicenter Comparative Clinical Trial of Lamotrigine or Carbamazepine for Cognitive Function as Initial Monotherapy in Adult Untreated Epilepsies
Brief Title: Lamotrigine Cognitive Function Study in Adult Untreated Epilepsies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korean Epilepsy Society (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Korean Epilepsy Society Chairman, Korean Epilepsy Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 106172
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; lamotrigine; cognitive function
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): lamotrigine
  Interventions: Drug: lamotrigine (Lamictal)
- 2 (Active Comparator): carbamazepine
  Interventions: Drug: Carbamazepine (Tegretol)

INTERVENTIONS:
Drug: lamotrigine (Lamictal) — lamotrigine: titration for 8 weeks (25 mg~200 mg per 2 weeks) and maintenance for 40 weeks (200 mg)
  Other Names: lamictal
  Arms: 1
Drug: Carbamazepine (Tegretol) — Carbamazepine: titration for 8 weeks (100 mg~600 mg) and maintenance for 40 weeks (600 mg)
  Other Names: Tegretol
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effect of anti-epileptic drugs' (AEDs) long-term treatment on cognitive function. This study is an open-label, randomized, multicenter comparative trial of lamotrigine versus carbamazepine. The planned enrollment is 100 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age : 16~60
* Seizure type was defined by MRI etc.
* Had more than 2 unprovoked seizures or 1 seizure with clear evidence for epilepsy (ex. positive in EEG or brain imaging)
* Need AED therapy and no AED medication for previous 1 year (exclude emergency medication for less than 2 weeks, baseline 4 weeks before)
* Is not pregnant by pregnancy test and is using contraceptive method
* Can report seizure diary by him/herself or his/her sick nurse
* Agreed to trial by written consent

Exclusion Criteria:

* Follow-up loss
* Canceled agreement
* Added other medication due to aggravated disease in 24 weeks
* Diagnosed as IGE
* Has progressive CNS disease by MRI or EEG
* Has serious systemic or psychological disease
* Under IQ 70
* Baseline lad data abnormality: Creatinine 2.0mg/dl or GOT/GPT 2 times higher than normal
* Abuse experience on alcohol or drugs
* Has experience on serious adverse event of any drug
* Previous experience on lamotrigine or carbamazepine
* Not suitable patients by investigator (uncooperative)
* Other reason which may interrupt the trial

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 121 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To define the superiority of Lamictal in cognitive function comparing to carbamazepine in newly diagnosed adult partial epilepsy patients | 48 weeks

SECONDARY OUTCOMES:
Seizure outcome and tolerability | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Ahm Lee, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea